CLINICAL TRIAL: NCT04673214
Title: Prognostic Modification in Patients With COVID-19 Under Early Intervention Treatment at U.M.F 13 and U.M.F 20
Brief Title: Evaluation of Prognostic Modification in COVID-19 Patients in Early Intervention Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilberto Cruz Arteaga (Other Government)
Collaborators: Coordinación de Investigación en Salud, Mexico (Other Government)
Responsible Party: Sponsor-Investigator, Gilberto Cruz Arteaga, Clinical Coordinator of Health Education and Research, Coordinación de Investigación en Salud, Mexico
Organization: Coordinación de Investigación en Salud, Mexico (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R-2020-785-176
Record Dates: First submitted 2020-12-16; First posted 2020-12-17 (Actual); Results first posted 2021-08-16 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Azithromycin; Ivermectin; Acetaminophen

STUDY DESIGN:
Intervention Model Description: Two groups of patients with COVID-19 will be integrated, a Group A taking the following medications: Paracetamol 500 mg orally 1 tablet every 8 hours for 3 days in case of fever equal to or greater than 38.3 ° C, Azithromycin tablets of 500 mg will take 1 single dose tablet the first day and then half a tablet (250 mg) orally every 24 for 4 days, Ivermectin tablets of 200mcg which will be calculated according to your weight and dose, it will be every 24 hours for 2 days and Rivaroxaban 10 mg tablets will take 1 every 24 hours for 10 days and a Group B will take Paracetamol 500 mg orally 1 tablet every 8 hours for 3 days in case of fever equal to or greater than 38.3 ° C, Azithromycin tablets of 500 mg will take 1 single dose tablet on the first day and then half a tablet orally every 24 hours for 4 days and Rivaroxaban 10 mg tablets will take 1 every 24 hours for 10 days.
Who Masked: Participant
Masking Description: For the conformation of the groups, random numbers generated by lottery will be used in which the patient will take a piece of paper as he arrives and will have the number of the group to which he will be assigned. With a type of block randomization, A (Azithromycin, paracetamol, Ivermectin, and Ribaroxaban) and B (paracetamol, Azithromycin, and Ribaroxaban).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Triple therapy (Experimental): Paracetamol 500 mg orally 1 tablet every 8 hours for 3 days in case of fever equal to or greater than 38.3 ° C, Azithromycin 500 mg tablets will take 1 tablet single dose the first day and then half tablet (250 mg) orally every 24 for 4 days, Ivermectin tablets of 200mcg which will be calculated according to your weight and dose, will be every 24 hours for 2 days and Rivaroxaban tablets of 10 mg will take 1 every 24 hours for 10 days
  Interventions: Drug: Azithromycin / Ivermectin / Ribaroxaban / Paracetamol
- Double therapy (Active Comparator): Paracetamol 500 mg orally 1 tablet every 8 hours for 3 days in case of fever equal to or greater than 38.3 ° C, Azithromycin 500 mg tablets will take 1 tablet single dose the first day and then half a tablet orally every 24 for 4 days and Rivaroxaban 10 mg tablets will take 1 every 24 hours for 10 days.
  Interventions: Drug: Azithromycin / Ribaroxaban / Paracetamol

INTERVENTIONS:
Drug: Azithromycin / Ivermectin / Ribaroxaban / Paracetamol — In the patient with the presence of COVID-19 confirmed by the PCR-COVID-19 positive test, the drug is randomly assigned to belong to group A of Azithromycin / Ivermectin / Ribaroxaban / Paracetamol to be followed for 14 days by video call (approximately 15 to 20 min per day) to the patient and the presence or absence of clinical symptoms, adverse reactions being recorded daily
  Other Names: with Ivermectin
  Arms: Triple therapy
Drug: Azithromycin / Ribaroxaban / Paracetamol — In the patient with the presence of COVID-19 confirmed by the PCR-COVID-19 positive test, the drug is randomly assigned to belong to group B of Azithromycin / Ribaroxaban / Paracetamol, to be followed for 14 days by video call (approximately 15 to 20 min per day) to the patient and the presence or absence of clinical symptoms, adverse reactions being recorded daily
  Other Names: without Ivermectin
  Arms: Double therapy

SUMMARY:
The present study is designed for patients with mild COVID-19 phase, to demonstrate if there is a modification in the clinical evolution greater than or equal to 25% in their symptoms, implemented in two groups of patients under an early intervention treatment, a group ( A) will receive Azithromycin / Ivermectin / Ribaroxaban / Paracetamol and another group (B) will receive Azithromycin / Ribaroxaban / Paracetamol followed for 14 days followed by video call

DETAILED DESCRIPTION:
Coronavirus disease (COVID-19) is caused by SARS-COV2 and represents the causative agent of a potential fatal disease generating a global public health problem. Person-to-person transmission of COVID-19 infection led to the isolation of patients who subsequently received a variety of treatments. Ivermectin treatment for safety is approved for human use by the FDA in parasitic and skin infections. Studies report the therapeutic safety of Ivermectin in humans with COVID-19, describing a 6.1-fold decrease in lethality compared to patients who did not use Ivermectin (1.4 vs. 8.5%, p <0.0001). In this sense, the WHO and PAHO encourage the use of unproven therapies in the context of a randomized clinical trial (RCT). Anticoagulants have reported up to 20% in the reduction of mortality (heparin), Ribaroxaban is effective with the inhibition of PAR1 / PAR2 / PAR4 receptors through the blocking of Factor Xa and the formation of thrombin, having anti-inflammatory effects, decreasing arteriosclerosis and platelet aggregation. There is a Telemedicine working method implemented by the OOAD of the North Federal District, which detects early signs and symptoms of possible complications and offers an early intervention treatment policy for first-level care beneficiaries. Under this method, a quasi-experimental study showed that there is a modification in the frequency of recovered patients of 80-90% in patients diagnosed with COVID-19 after an early intervention treatment with paracetamol, Ivermectin, Azithromycin, Ribaroxaban in patients with COVID -19 from UMF 13 during the period of July-August 2020. Therefore, it is necessary to carry out a randomized clinical trial to confirm this assertion.

Objective: To evaluate the percentage of patients with a diagnosis of COVID-19 who modify their clinical evolution under a comparative treatment of early intervention in beneficiaries of the U.M.F 13 and U.M.F 20 of the I.M.S.S., during the period of December 2020-January 2021.

Material and Methods: A randomized, single-blind, prospective, longitudinal and open experimental study in 62 patients with COVID-19 from UMF No. 13 and No. 20 from November to December 2020. Including 31 patients in group A (Azithromycin / Ivermectin / Ribaroxaban / Paracetamol) and 31 patients in group B (Azithromycin / Ribaroxaban / Paracetamol). With inclusion criteria over 18 years of age, have type 2 diabetes mellitus, Systemic Arterial Hypertension, Obesity or overweight, PCR confirmation of COVID-19. For the video call, the Family Medicine Units have Electronic Equipment Installation for Internet use. Exclusion criteria are patients with severe COVID-19 (they deserve immediate referral to second level of care, hospital). Elimination criteria are Prior informed consent, medication is given randomly to a COVID-19 patient, a follow-up video call will be made at home for 14 days, recording sex, age, education, date of disease onset, taking laboratories (hematic biometry, C-reactive protein, D-dimer, Ferritin, prothrombin time, thromboplastin time, lactic dehydrogenase) taken at the onset of the disease, taking as an outcome variable the modification of the clinical course (clinical symptoms such as headache, cough, fever, conjunctivitis , myalgias, arthralgias, rhinorrhea, odynophagia, anosmia, chest pain, dyspnea) when granting treatment in groups A and B.. Statistical differences will be evaluated using the Mann-Whitney U test with a power of 90% and a type I error rate of 1% for the variable of modification of the clinical course in treatment groups A and B. analysis will be performed in SPSS version 21.

ELIGIBILITY:
Inclusion Criteria:

* Patients Eligible for Family Medicine Unit No.20 and Family Medicine Unit No.13 belonging to the North DF of the IMSS.
* Male and female patients
* Patients over 18 years of age.
* Patients with compliance with the operational definition COVID-19 and confirmatory test of P.C.R. positive within the first days of the illness (that are evaluated in first level of medical attention).
* Patients with comorbidities such as Type 2 Diabetes Mellitus, Systemic Arterial Hypertension, Overweight or Obesity.
* That they agree to sign an informed consent

  - Related to Video Call:
* That the Family Medicine Unit No.20 and the Family Medicine Unit No.13 belonging to the North DF of the IMSS have the Installation of Electronic Equipment for Internet use

Exclusion Criteria:

* Severe COVID-19 patients (Ameriten sent immediately to second level of care, hospital) Patients with any Personal Pathological History of Hematological Diseases. • Patients allergic to macrolides (Azithromycin) and Ivermectin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2020-12-16 (Actual); Primary Completion 2021-02-25 (Actual); Study Completion 2021-02-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GILBERTO CR ARTEAGA, specialist, Principal Investigator — MEXICAN SOCIAL SECURITY INSTITUTE
Locations (1):
- Alma Italia Guerrero Martinez, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No
SHARED VIA EMAIL IF OTHER RESEARCHERS REQUIRE IT

REFERENCES:
- [Background] Gautret P, Lagier JC, Parola P, Hoang VT, Meddeb L, Mailhe M, Doudier B, Courjon J, Giordanengo V, Vieira VE, Tissot Dupont H, Honore S, Colson P, Chabriere E, La Scola B, Rolain JM, Brouqui P, Raoult D. RETRACTED: Hydroxychloroquine and azithromycin as a treatment of COVID-19: results of an open-label non-randomized clinical trial. Int J Antimicrob Agents. 2020 Jul;56(1):105949. doi: 10.1016/j.ijantimicag.2020.105949. Epub 2020 Mar 20. PMID 32205204
- [Background] Becattini C, Pace U, Rondelli F, Delrio P, Ceccarelli G, Boncompagni M, Graziosi L, Visona A, Chiari D, Avruscio G, Frasson S, Gussoni G, Biancafarina A, Camporese G, Donini A, Bucci AF, Agnelli G. Rivaroxaban for extended antithrombotic prophylaxis after laparoscopic surgery for colorectal cancer. Design of the PRO-LAPS II STUDY. Eur J Intern Med. 2020 Feb;72:53-59. doi: 10.1016/j.ejim.2019.11.015. Epub 2019 Dec 7. PMID 31818628
- [Background] Khorana AA, Soff GA, Kakkar AK, Vadhan-Raj S, Riess H, Wun T, Streiff MB, Garcia DA, Liebman HA, Belani CP, O'Reilly EM, Patel JN, Yimer HA, Wildgoose P, Burton P, Vijapurkar U, Kaul S, Eikelboom J, McBane R, Bauer KA, Kuderer NM, Lyman GH; CASSINI Investigators. Rivaroxaban for Thromboprophylaxis in High-Risk Ambulatory Patients with Cancer. N Engl J Med. 2019 Feb 21;380(8):720-728. doi: 10.1056/NEJMoa1814630. PMID 30786186
- [Background] Dugina TN, Kiseleva EV, Chistov IV, Umarova BA, Strukova SM. Receptors of the PAR family as a link between blood coagulation and inflammation. Biochemistry (Mosc). 2002 Jan;67(1):65-74. doi: 10.1023/a:1013952114485. PMID 11841341
- [Background] Choudhary R, Sharma AK. Potential use of hydroxychloroquine, ivermectin and azithromycin drugs in fighting COVID-19: trends, scope and relevance. New Microbes New Infect. 2020 Apr 22;35:100684. doi: 10.1016/j.nmni.2020.100684. eCollection 2020 May. PMID 32322397
- [Background] Arshad U, Pertinez H, Box H, Tatham L, Rajoli RKR, Curley P, Neary M, Sharp J, Liptrott NJ, Valentijn A, David C, Rannard SP, O'Neill PM, Aljayyoussi G, Pennington SH, Ward SA, Hill A, Back DJ, Khoo SH, Bray PG, Biagini GA, Owen A. Prioritization of Anti-SARS-Cov-2 Drug Repurposing Opportunities Based on Plasma and Target Site Concentrations Derived from their Established Human Pharmacokinetics. Clin Pharmacol Ther. 2020 Oct;108(4):775-790. doi: 10.1002/cpt.1909. Epub 2020 Jun 14. PMID 32438446
- See also: Hydroxychloroquine and azithromycin as a treatment of COVID-19: results of an open-label non-randomized clinical trial — https://doi.org/10.1016/j.ijantimicag.2020.105949
- See also: Effectiveness of Ivermectin as add-on Therapy in COVID-19 Management — https://clinicaltrials.gov/ct2/show/results/NCT04343092?term=NCT04343092&draw=2&rank=1&view=results

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment begins on December 16, 2020 in the Family Medicine Unit No.13 and in the Family Medicine Unit No.20 of the Mexican Institute of Social Security.
Pre-assignment Details: There were no excluded patients.
Groups:
- Triple Therapy: 65 triple therapy patients received the assigned intervention with Azithromycin tablets 500 mg 1 tablet in a single dose the first day and then half a tablet (250 mg) orally every 24 4 days, ivermectin tablets of 200 mcg calculated according to your weight and dose, will be every 24 hours for 2 days and Rivaroxaban 10 mg tablets take 1 every 24 hours for 10 days and Paracetamol 500 mg orally 1 tablet every 8 hours for 3 days in case of fever equal to or greater than 38.3 ° C.
- Double Therapy: 46 double therapy patients received the assigned intervention with Azithromycin 500 mg tablets 1 single dose tablet on the first day and then half a tablet (250 mg) orally every 24 4 days and rivaroxaban 10 mg tablets take 1 every 24 hours for 10 days with Paracetamol 500 mg orally 1 tablet every 8 hours for 3 days in case of fever equal to or greater than 38.3 ° C.
Period: Overall Study
Arm/Group | Triple Therapy | Double Therapy
Started | 67 | 47
Lost to Follow up | 2 (These patients were discontinued, given in the first days of their follow-up by video call, they presented major symptoms such as dyspnea of movement, dyspnea at rest, and chest pain; Following the protocol's follow-up criteria, patients were informed of their clinical care at the hospital level immediately, and the protocol was no longer followed. Subsequently, when capturing information in the data analysis, the clinical status of the patients is searched, registering their death.) | 1 (This patient was stopped being followed up in the first days of his follow-up by video call. He presented major symptoms such as dyspnea of movement, dyspnea at rest, and chest pain; With the follow-up criteria of the protocol, the patient was informed of their clinical care at the hospital level immediately, and the protocol was no longer followed. Subsequently, when capturing information in the data analysis, the clinical status of the patient is searched, registering death.)
Completed (Analyzed) | 65 | 46
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Population: Assuming a 25% efficacy in modifying the clinical course (COVID-19 mild phase symptoms) of patients with COVID-19 under a comparative treatment for 14 days followed by video call, with a power of 90%, type I error rate 1% and loss to follow-up 20%; A total of 62 patients was calculated, however due to the availability of medication, it was recalculated to 111 patients, that is, 65 cases in the triple therapy group and 46 in the double therapy group would be necessary for the analysis.
Groups:
- Double Therapy: The following medications were taken for this group: Azithromycin 500 mg tablets take 1 single dose tablet the first day and then half a tablet (250 mg) orally every 24 for 4 days; Rivaroxaban 10 mg tablets take 1 every 24 hours for 10 days; Paracetamol 500 mg orally take 1 tablet every 8 hours for 3 days in case of fever equal to or greater than 38.3 ° C.
- Triple Therapy: The following medications were taken for this group: Azithromycin 500 mg tablets take 1 single dose tablet the first day and then half a tablet (250 mg) orally every 24 for 4 days; Ivermectin 6 mg tablets take as follows 2 TABLETS <80 KG orally, 3 TABLETS between 80-110 kg orally, 4 TABLETS> 110kg orally, every 24 hours for 2 days; Rivaroxaban 10 mg tablets take 1 every 24 hours for 10 days; Paracetamol 500 mg orally take 1 tablet every 8 hours for 3 days in case of fever equal to or greater than 38.3 ° C.
- Total: Total of all reporting groups
Arm/Group | Double Therapy | Triple Therapy | Total
Number analyzed (Participants) | 46 | 65 | 111
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 46 | 61 | 107
  >=65 years | 0 | 4 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 34 | 58
  Male | 22 | 31 | 53
Race/Ethnicity, Customized [Number; unit: participants]
  Mestizo Mexicans | 46 | 65 | 111
Region of Enrollment [Count of Participants; unit: Participants]
  Mexico | 46 | 65 | 111
Age [Count of Participants; unit: Participants]
  21-30 years | 8 | 6 | 14
  31-40 years | 12 | 17 | 29
  41-50 years | 14 | 22 | 36
  51-60 years | 7 | 8 | 15
  61-70 years | 5 | 8 | 13
  ≥ 71 years | 0 | 4 | 4
Occupation [Count of Participants; unit: Participants]
  Part time | 2 | 11 | 13
  Full time | 41 | 40 | 81
  Housewife | 1 | 4 | 5
  Pensioner | 2 | 9 | 11
  Unemployed | 0 | 1 | 1
Civil Status [Count of Participants; unit: Participants]
  Single | 12 | 13 | 25
  Married | 25 | 44 | 69
  Widower | 1 | 1 | 2
  Free Union | 7 | 5 | 12
  Divorced | 1 | 2 | 3
Education [Count of Participants; unit: Participants]
  Primary | 2 | 1 | 3
  High school | 3 | 9 | 12
  Preparatory | 13 | 9 | 22
  Technical career | 4 | 4 | 8
  Degree | 21 | 32 | 53
  Others | 3 | 10 | 13

OUTCOME MEASURES:

1. Primary Outcome: Average Days in COVID-19 Symptoms by Type of Therapy in the UMF 20 and UMF 13 of the IMSS.
Description: Statistical differences were evaluated using Student's t test for quantitative variables. In relation to the presence of the number of days with clinical symptoms of COVID-19 by double therapy vs. triple therapy.
Time Frame: 14 days
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: days
Arm/Group | DOUBLE THERAPY | TRIPLE THERAPY
Number analyzed (Participants) | 46 | 65
days
  Cough | 7 (5.4) | 7 (5.6)
  Fever | 2 (3.4) | 2 (3.2)
  Headache | 6 (5.2) | 5 (4.9)
  Rhinorrhea | 3 (4.8) | 3 (4.3)
  Odynophagia | 5 (4.8) | 5 (5.4)
  Diarrhea | 2 (4) | 1 (2.2)
  Myalgia | 6 (5.6) | 5 (5)
  Anosmia | 5 (5.8) | 6 (5.9)
  Conjunctivitis | 2 (4.1) | 1 (2.9)
  Chest pain | 5 (5.6) | 4 (4.8)
  Dyspnea of movement | 2 (4.1) | 2 (3.9)
  Dysnea at rest | 1 (3.3) | 2 (3.6)
  Major symptoms | 5 (3.1) | 5 (3.4)
  Minor symptoms | 3 (2.7) | 3 (2.5)
  treatment start day | 4 (1.9) | 4 (1.6)
Statistical Analysis 1: Comparison: DOUBLE THERAPY vs TRIPLE THERAPY; Null Hypothesis: There will be no modification in the clinical evolution ≥ 25% of patients diagnosed with COVID-19 under an early intervention treatment with Azithromycin / Ivermectin / Ribaroxaban / Paracetamol vs. Azithromycin / Ribaroxaban / Paracetamol for 14 days followed by video call from U.M.F 13 and U.M.F 20 from I.M.S.S., during the period of December 2020- February 2021, with a power of 90%, type I error rate 1% and loss to follow-up 20%; Test type: Superiority — The null hypothesis for the modification in the clinical evolution of the conjunctivitis sign in patients diagnosed with COVID-19 under early intervention treatment with Azithromycin / Ribaroxaban / Paracetamol for 14 days followed by video call is rejected; p = 0.05, Chi-squared — Presence of a p <0.05 as significant in the comparison of treatment with clinical symptoms
Statistical Analysis 2: Comparison: DOUBLE THERAPY vs TRIPLE THERAPY; Assuming a difference of 2 days in the modification of the clinical course (symptoms of fever, cough, headache, myalgia, odynophagia, anosmia, rhinorrhea, arthralgia, chest pain, dyspnea, conjunctivitis) of patients diagnosed with COVID-19 in early intervention treatment vs. therapeutic failure, for 14 days followed by video call, with a power of 90%, a type I error rate of 1% and a loss to follow-up of the twenty%; Test type: Superiority — The null hypothesis is rejected with a difference of 2 days in the modification of the clinical evolution (symptoms of fever, cough, headache, myalgia, odynophagia, anosmia, rhinorrhea, arthralgia, chest pain, dyspnea, conjunctivitis) of patients diagnosed with COVID -19 in early intervention treatment. vs. therapeutic failure, for 14 days followed by video call, with a power of 90%, a type I error rate of 1% and a loss to follow-up of 20%; p = 0.05, t-test, 2 sided

2. Primary Outcome: Crosstabulated Outcome in Modification of the Evolution Clinical vs Fails Therapeutic by Type of Treatment in Patients With COVID-19 UMF 13 and UMF 20 of the IMSS
Description: Statistical differences between clinical evolution vs therapeutic failure by type of treatment were evaluated using Pearson's Chi-square test as categorical variables.
Time Frame: 14 days
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Double Therapy | Triple Therapy
Number analyzed (Participants) | 46 | 65
Participants
  Number of Participants with Improvement in Clinical Evaluation | 44 | 59
  Number of Participants with Therapeutic Failure | 2 | 6
Statistical Analysis 1: Comparison: Double Therapy vs Triple Therapy; Assuming a difference in the percentage of effectiveness in the clinical modification and therapeutic failure of patients diagnosed with COVID-19 under treatment with Azithromycin / Ivermectin / Ribaroxaban / Paracetamol vs. Azithromycin / Ribaroxaban / Paracetamol followed for 14 days followed by video call, with a power of 90%, a type I error rate of 1% and a loss to follow-up of 20%; Test type: Superiority — Assuming a difference in the percentage of effectiveness in the clinical modification and therapeutic failure of patients diagnosed with the outcome of improvement in the Modification of the clinical evolution of the symptoms of patients with COVID-19 using double therapy was reported 95.7% (n = 44) Vs. triple therapy 90.8% (n = 59) and therapeutic failure 4.3% (n = 2) vs. 9.2% (n = 6), respectively; p = 0.05, Chi-squared — Presence of a p <0.05 as significant in the comparison of treatment with clinical symptoms the clinical modification and therapeutic failure of patients diagnosed with COVID-19

3. Other Pre Specified Outcome: Average Days of COVID-19 Symptoms Under Treatment of Early Intervention Due to Outcome in UMF 13 and 20 of the IMSS
Description: Statistical differences were evaluated using Student's t test for quantitative variables. The average duration of days with clinical symptoms of COVID-19 under early intervention treatment by outcome in the improvement of the modification of the clinical evolution of symptoms vs. therapeutic failure.
Time Frame: 14 days
Population: Assuming a difference in days of effectiveness in clinical modification and therapeutic failure of patients diagnosed with COVID-19 in treatment with Azithromycin / Ivermectin / Ribaroxaban / Paracetamol vs. Azithromycin / Ribaroxaban / Paracetamol followed for 14 days followed by video call, with a potency 90%, a Type I error rate of 1%, and a loss to follow-up of 20%
Measure: Mean (Standard Deviation); unit: Days
Groups:
- Modification of Evolution Clinic: Improvement of the clinical health conditions of symptoms such as headache, cough, fever, conjunctivitis, myalgia, arthralgia, rhinorrhea, odynophagia, anosmia, chest pain, dyspnea after the administration of the dual therapy of Azithromycin / Ribaroxaban / Paracetamol and the Azithromycin / Ivermectin / Ribaroxaban / Paracetamol triple therapy in patients with mild Covid-19 clinical phase performed by video call monitoring lasting 15-20 minutes for 14 days.
- Therapeutic Failure: Lack of efficacy after the administration of Azithromycin / Ribaroxaban / Paracetamol dual therapy and Azithromycin / Ivermectin / Ribaroxaban / Paracetamol triple therapy in the registry of clinical health conditions of symptoms such as headache, cough, fever, conjunctivitis, myalgia, arthralgia , rhinorrhea, odynophagia, anosmia, chest pain, dyspnea, of patients with mild clinical phase Covid-19 performed by monitoring with a duration of 15-20 minutes during 14 days of follow-up.
Arm/Group | Modification of Evolution Clinic | Therapeutic Failure
Number analyzed (Participants) | 103 | 8
Days
  Cough | 7 (5.6) | 4 (3.3)
  Fever | 2 (3.3) | 1 (1.7)
  Headache | 6 (5) | 2 (2)
  Rhinorrhea | 4 (4.6) | 1 (1.4)
  Odynophagia | 5 (5.2) | 2 (3.2)
  Diarrhea | 2 (3.2) | 1 (2.1)
  Myalgia | 6 (5.4) | 5 (2)
  Anosmia | 6 (6) | 2 (2.3)
  Conjunctivitis | 1 (3.6) | 1 (1.4)
  Chest Pain | 4 (5.2) | 1 (1.5)
  Dyspnea of movement | 2 (4.1) | 3 (2.9)
  Dyspnea at Rest | 1 (3.5) | 3 (2.9)
  Major Symptoms | 5 (3.3) | 2 (1.5)
  Minor Symptoms | 3 (2.6) | 2 (1.2)
Statistical Analysis 1: Comparison: Modification of Evolution Clinic vs Therapeutic Failure; Assuming a difference in days of effectiveness in clinical modification and therapeutic failure of patients diagnosed with COVID-19 in treatment with Azithromycin / Ivermectin / Ribaroxaban / Paracetamol vs. Azithromycin / Ribaroxaban / Paracetamol followed for 14 days followed by video call, with a potency 90%, a Type I error rate of 1%, and a loss to follow-up of 20%; Test type: Superiority — The null hypothesis is rejected with a mean duration of 2 days with clinical symptoms of COVID-19 in early intervention treatment as a result of improving the modification of the clinical evolution of symptoms vs therapeutic failure; p = 0.05, t-test, 2 sided

4. Other Pre Specified Outcome: Number of Participants Who Were Alive and Had COVID-19 Symptoms by Type of Therapy During a 14-day Follow-up
Description: Survival analysis. The time it takes for 50% of COVID-19 patients to improve symptoms during a 14-day follow-up with dual therapy vs. triple therapy
Time Frame: 14 days
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Double Therapy | Triple Therapy
Number analyzed (Participants) | 46 | 65
Participants
  Cought | 16 | 26
  Fever | 10 | 7
  Headache | 6 | 7
  Odynophagia | 26 | 35
  Rhinorrhea | 17 | 16
  Anosmia | 34 | 33
  Conjunctivitis | 13 | 8
  Diarrhea | 8 | 11
  Myalgia | 23 | 35
  Chest pain | 25 | 33
  Dyspnea of movement | 14 | 18
  Dyspnea at rest | 9 | 16
Statistical Analysis 1: Comparison: Double Therapy vs Triple Therapy; Assuming a 25% efficacy in modifying the clinical course (COVID-19 mild phase symptoms) of patients with COVID-19 under a comparative treatment for 14 days followed by video call, with a power of 90%, type I error rate 1% and loss to follow-up 20%; Test type: Superiority — A total of 62 patients was calculated, however due to the availability of medication, it was recalculated to 111 patients, that is, 65 cases in the triple therapy group and 46 in the double therapy group would be necessary for the analysis; p = 0.05, Wilcoxon (Gehan) statistical test

ADVERSE EVENTS:
Time Frame: Adverse event data was collected was 14 days.
Description: No presence of serious adverse events
Groups:
- Dual Therapy Adverse Event: Record of adverse reactions of Blood and lymphatic system disorders, Heartdisorders, Ear and labyrinth disorders,Gastrointestinal disorders and Musculoskeletal and connective tissue disorders with the following medications were taken for this group: Azithromycin 500 mg tablets take 1 single dose tablet the first day and then half a tablet (250 mg) orally every 24 for 4 days; Rivaroxaban 10 mg tablets take 1 every 24 hours for 10 days; Paracetamol 500 mg orally take 1 tablet every 8 hours for 3 days in case of fever equal to or greater than 38.3 ° C.
- Adverse Event Triple Therapy: Record of adverse reactions of Blood and lymphatic system disorders, Heartdisorders, Ear and labyrinth disorders,Gastrointestinal disorders and Musculoskeletal and connective tissue disorders with the following medications were taken for this group: Azithromycin 500 mg tablets take 1 single dose tablet the first day and then half a tablet (250 mg) orally every 24 for 4 days; Ivermectin 6 mg tablets take as follows 2 TABLETS <80 KG orally, 3 TABLETS between 80-110 kg orally, 4 TABLETS> 110kg orally, every 24 hours for 2 days; Rivaroxaban 10 mg tablets take 1 every 24 hours for 10 days; Paracetamol 500 mg orally take 1 tablet every 8 hours for 3 days in case of fever equal to or greater than 38.3 ° C.
Arm/Group | Dual Therapy Adverse Event | Adverse Event Triple Therapy
All-Cause Mortality (participants affected / at risk) | 1/46 | 2/65
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/65
Other Adverse Events (participants affected / at risk) | 39/46 | 49/65
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dual Therapy Adverse Event (N=46) | Adverse Event Triple Therapy (N=65)
asthenia (Skin and subcutaneous tissue disorders) | 24 (24) | 18 (18) — Symptom presented in patients without causing without requiring immediate medical attention or subsequent clinical follow-up
Palpitations (Cardiac disorders) | 4 (4) | 5 (5) — Symptom presented in patients without causing without requiring immediate medical attention or subsequent clinical follow-up.
Tinnitus (Ear and labyrinth disorders) | 6 (6) | 10 (10) — Symptom presented in patients without causing without requiring immediate medical attention or subsequent clinical follow-up.
Nausea (Gastrointestinal disorders) | 9 (9) | 18 (18) — Symptom presented in patients without causing without requiring immediate medical attention or subsequent clinical follow-up.
Ecchymosis (Blood and lymphatic system disorders) | 2 (2) | 2 (2) — Symptom presented in patients without causing without requiring immediate medical attention or subsequent clinical follow-up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-12-11): https://cdn.clinicaltrials.gov/large-docs/14/NCT04673214/Prot_SAP_000.pdf
  • Informed Consent Form (2020-12-11): https://cdn.clinicaltrials.gov/large-docs/14/NCT04673214/ICF_001.pdf